CLINICAL TRIAL: NCT04585854
Title: Effect of Caffeine on Myocardial Oxygenation
Acronym: Coffee-O2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-01876
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Caffeine
Keywords: CMR; Myocardial oxygenation; Myocardial Function; Coffee
MeSH Terms: interventions — Caffeine; Coffee

STUDY DESIGN:
Intervention Model Description: Controlled before-after comparison
Masking Description: Blinded image analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Other): Control population who will undergo two cardiovascular magnetic resonance exams: one at rest and one after drinking caffeine.
  Interventions: Other: Caffeine

INTERVENTIONS:
Other: Caffeine — Consumption of 3 shots of espresso
  Other Names: Coffee

SUMMARY:
The purpose of this study is to investigate the impact of caffeine on myocardial oxygenation and other cardiovascular magnetic resonance parameters in healthy controls.

DETAILED DESCRIPTION:
Caffeine is presumed to create a confounder with diagnostic imaging. The vasodilatory capacity is considered a key measure for the detection of significant coronary disease with stenosed epicardial arterial conduit vessels and overall microvascular function, including endothelial dysfunction. Twenty nine healthy controls will undergo a baseline cardiovascular magnetic resonance (CMR) exam. Afterwards, participants will consume coffee in the presence of study personnel. This will consist of 3 espresso shots, which will be consumed within 15 minutes. Approximately 2h after coffee consumption the CMR exam will be repeated. The goal will be to investigate the impact of caffeine on myocardial features. In particular the effect on the myocardial oxygenation response to vasodilating and vasoconstricting stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent, documented by signature
* Aged 18 to 45

Exclusion Criteria:

* MRI Contraindications following current institutional guidelines at the time of the CMR exam
* Knowledge or suspicion of pregnancy (verified with a pregnancy test).
* Consumption of caffeine 12h prior to the baseline CMR exam (outside of the study protocol).
* Known cardiovascular disease, diabetes, severe respiratory disease, obstructive sleep apnea syndrome, chemotherapy and radiation treatment, cerebrovascular and occlusive peripheral vascular disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Difference in myocardial oxygenation responses | Through study completion up to 5 hours, before and after caffeine
  Percent (%) Measure of oxygenation-sensitive signal change measured by CMR

SECONDARY OUTCOMES:
Difference in ejection fraction | Through study completion up to 5 hours, before and after caffeine
  Percent (%), measured by CMR
Difference in cardiac index | Through study completion up to 5 hours, before and after caffeine
  L/min/m2, measured by CMR
Difference in myocardial peak strain | Through study completion up to 5 hours, before and after caffeine
  Percent (%), a measure of systolic function (shortening and thickening) of the myocardium measured by CMR
Difference in myocardial time to peak strain | Through study completion up to 5 hours, before and after caffeine
  Milliseconds (ms), measured by CMR
Difference in myocardial strain rate | Through study completion up to 5 hours, before and after caffeine
  Change in strain over time (/second), measured by CMR
Difference in myocardial parametric mapping | Through study completion up to 5 hours, before and after caffeine
  Milliseconds (ms), measured by CMR
Difference in 4D blood flow | Through study completion up to 5 hours, before and after caffeine
  Percent, measured by CMR
Difference in rate pressure product | Through study completion up to 5 hours, before and after caffeine
  Blood pressure * heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Dominik P Guensch, MD, Principal Investigator — Bern University Hospital, Inselspital
Locations (1):
- Bern University Hospital, Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Fischer K, Yamaji K, Luescher S, Ueki Y, Jung B, von Tengg-Kobligk H, Windecker S, Friedrich MG, Eberle B, Guensch DP. Feasibility of cardiovascular magnetic resonance to detect oxygenation deficits in patients with multi-vessel coronary artery disease triggered by breathing maneuvers. J Cardiovasc Magn Reson. 2018 May 7;20(1):31. doi: 10.1186/s12968-018-0446-y. PMID 29730991
- [Background] van Dijk R, Ties D, Kuijpers D, van der Harst P, Oudkerk M. Effects of Caffeine on Myocardial Blood Flow: A Systematic Review. Nutrients. 2018 Aug 13;10(8):1083. doi: 10.3390/nu10081083. PMID 30104545
- [Background] Kuijpers D, Prakken NH, Vliegenthart R, van Dijkman PR, van der Harst P, Oudkerk M. Caffeine intake inverts the effect of adenosine on myocardial perfusion during stress as measured by T1 mapping. Int J Cardiovasc Imaging. 2016 Oct;32(10):1545-53. doi: 10.1007/s10554-016-0949-2. Epub 2016 Jul 29. PMID 27473274